CLINICAL TRIAL: NCT07109388
Title: Comparison of Pericapsular Nerve Group (PENG) Block With a Combined Femoral, Sciatic, Lateral Femoral Cutaneous Nerve Block for Postoperative Analgesia in Secondary Total Hip Arthroplasty.
Brief Title: Comparison of Pericapsular Nerve Group (PENG) Block With a Combined Femoral, Sciatic, Lateral Femoral Cutaneous Nerve Block for Postoperative Analgesia in Secondary Total Hip Arthroplasty; (REVPET)
Acronym: REVPET
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Vaudois (Other)
Responsible Party: Principal Investigator, Eric Albrecht, Prof. Dr. Med. Eric Albrecht, Associate Professor, University of Lausanne, Centre Hospitalier Universitaire Vaudois
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2025-00488
Record Dates: First submitted 2025-07-07; First posted 2025-08-07 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Hip Arthroplasty Replacement; Post Operative Analgesia; Post Operative Pain, Acute
Keywords: nerve block; postoperative pain; hip arthroplasty replacement
MeSH Terms: conditions — Pain, Postoperative | interventions — Dental Occlusion; Ropivacaine

STUDY DESIGN:
Intervention Model Description: This is a single-center, prospective, superiority, randomized, double-blind, parallel-group study.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PENG group (Experimental): Pericapsular nerve group block
  Interventions: Drug: Pericapsular nerve group (PENG) block with 0.75% ropivacaine guided by ultrasound
- Combined nerve block (Active Comparator): Combined femoral, sciatic, lateral femoral cutaneous nerve block
  Interventions: Drug: Femoral, sciatic and lateral femoral cutaneous nerve block with 0.375% ropivacaine

INTERVENTIONS:
Drug: Pericapsular nerve group (PENG) block with 0.75% ropivacaine guided by ultrasound — Participants in the PENG group will first receive a sham sciatic injection; the needle will be inserted into the subcutaneous tissue and 3 ml of 0.9% NaCl will be injected. They will then receive a PENG nerve block in the supine position. A low-frequency (2-5 MHz) curvilinear ultrasound probe (BK Ultrasound) will be used to identify the anterior inferior iliac spine, the pubic eminence, and the psoas tendon with its fascial plane. A 22-gauge, 50 mm needle (SonoPlex® Pajunk) will be inserted into the fascial plane to inject 20 ml of 0.75% ropivacaine (Fresenius Kabi).
  Other Names: PENG block
  Arms: PENG group
Drug: Femoral, sciatic and lateral femoral cutaneous nerve block with 0.375% ropivacaine — Participants in the combined group will first receive a sciatic nerve block performed with the patient in a semi-prone position, the lower limb flexed at 90° (hip and knee), elevated with a cushion placed between the legs. A straight line will be drawn between the greater trochanter and the ischial tuberosity. The sciatic nerve is located approximately at the midpoint of this line. Under ultrasound guidance, the ischial tuberosity will be identified medially, the greater trochanter laterally, the gluteus maximus muscle superficially beneath the adipose tissue, and the quadratus femoris muscle in depth. A 22-gauge, 50 mm needle will then be inserted into the fascial plane to inject 20 ml of 0.375% ropivacaine. The patient is then placed supine for femoral and lateral femoral cutaneous nerve blocks. 15 ml of local anaesthetics will be injected around the femoral nerve and 5 around the lateral femoral cutaneous nerve.
  Arms: Combined nerve block

SUMMARY:
The aim of this clinical trial is to compare the analgesic effect of a pericapsular nerve group (PENG) block with a combined femoral, sciatic, lateral femoral cutaneous nerve block for postoperative analgesia in patients scheduled for secondary total hip arthroplasty. The primary objective of this study is to compare postoperative pain management between the PENG block and the combined block (femoral, sciatic, lateral femoral cutaneous) by measuring postoperative morphine consumption in each of the two groups.

Participants will be randomized into two groups. Patients assigned to the PENG group will receive a PENG block with ropivacaine, followed by a sham (sciatic) block, and spinal anesthesia with isobaric bupivacaine. Patients assigned to the combined block group will receive femoral, sciatic, lateral femoral cutaneous nerve blocks with ropivacaine, followed by spinal anesthesia with isobaric bupivacaine.

DETAILED DESCRIPTION:
This is a single-center, prospective, superiority, randomized, double-blind, parallel-group study.

Patients will be randomized into two groups of 25 patients each, for a total enrollment plan of 50 patients. After written informed consent, patients will be allocated to one of the two groups according to a computer-generated randomization list.

The nerve blocks will be performed using ultrasound guidance.

During the surgery, 0.15 mg/kg of dexamethasone IV, 1 g paracetamol IV, 30 mg ketorolac IV, and 40 mg/kg magnesium IV will be given for postoperative analgesia.

In the PACU, pain management will be provided as needed with 2 mg of IV morphine at ten-minute intervals for pain scores >4. Once spinal motor block has resolved, the patients will be transferred to the surgical ward with a morphine patient-controlled analgesia (PCA) pump. The pump parameters will allow 2 mg boluses of morphine with a 10-minute lockout and a maximum dose of 40 mg in 4 hours.

Basal analgesia will be provided with paracetamol (1 g/6 h) and ibuprofen (400 mg/8 h). Ondansetron (4 mg IV) will be administered in case of nausea or vomiting.

A research assistant will conduct postoperative visits at 2 hours, 1 day, and 2 days postoperatively to record research data. Functional testing will be done on days 1 and 2 by physiotherapy personnel.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients
* ASA (American Society of Anaesthesiologists) I-III
* 18 years of age or older
* Patients scheduled for elective secundary hip arthroplasty
* Able to give written conformed consent autonomously

Exclusion Criteria:

* Refusal or inability to give consent
* Allergy to any of: ropivacaine, paracetamol, ibuprofen, ketorolac, morphine, ondansetron or dexamethasone
* Bleeding diathesis
* Neurological deficit of the operative side
* Existing preoperative opioid use
* Renal insufficiency (GFR<30ml/min according to the Cockroft-Gault formula)
* Hepatic insufficiency
* Morbid Obésity III

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-09-30 (Estimated); Primary Completion 2027-09-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
Cumulative postoperative morphine consumption at day 1 | Time Frame: 24 hours postoperatively
  Description: total consumption in mg

SECONDARY OUTCOMES:
Morphine consumption in the recovery room | from admission till discharge from the recovery room, up to 2 hours
  consumption in mg
PCA administered morphine consumption at day 2 | at day 2 postoperatively
  consumption in mg administered by PCA
Rest and dynamic pain scores | At 2 hours, day 1 and day 2 postoperatively
  Visual Analogue Scale(VAS), 0-10
Incidence of postoperative nausea and vomiting | at 2 hours, day 1 and day 2 postoperatively
  Presence of nausea or vomiting in the postoperative period
Incidence of pruritus | at 2 hours, day 1 and day 2 postoperatively
  Presence of pruritus in the postoperative period
Incidence of urinary retention requiring bladder catheterisation | from surgery till day 2 postoperatively
  Urinary retention requiring catheterisation
Duration of analgesia | from the time the study procedure is performed up to 36 hours after surgery
  Time between study procedure and the first dose of iv morphine
Operated limb quadriceps strength | At day 1 and day 2 postoperatively
  Medical Research Council Manual Muscle Testing scale, 0-5
Walking test | At day 1 and 2 postoperatively
  Maximum distance travelled (meters)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] She C, Liu H. The efficacy of pericapsular nerve group block for reducing pain and opioid consumption after total hip arthroplasty: a systematic review and meta-analysis. J Orthop Surg Res. 2024 Apr 8;19(1):229. doi: 10.1186/s13018-024-04707-x. PMID 38584259
- [Background] Newman JT, Briggs KK, McNamara SC, Philippon MJ. Outcomes After Revision Hip Arthroscopic Surgery in Adolescent Patients Compared With a Matched Cohort Undergoing Primary Arthroscopic Surgery. Am J Sports Med. 2016 Dec;44(12):3063-3069. doi: 10.1177/0363546516659656. Epub 2016 Aug 11. PMID 27514736
- [Background] Bohl DD, Samuel AM, Basques BA, Della Valle CJ, Levine BR, Grauer JN. How Much Do Adverse Event Rates Differ Between Primary and Revision Total Joint Arthroplasty? J Arthroplasty. 2016 Mar;31(3):596-602. doi: 10.1016/j.arth.2015.09.033. Epub 2015 Sep 28. PMID 26507527
- [Background] Mahomed NN, Barrett JA, Katz JN, Phillips CB, Losina E, Lew RA, Guadagnoli E, Harris WH, Poss R, Baron JA. Rates and outcomes of primary and revision total hip replacement in the United States medicare population. J Bone Joint Surg Am. 2003 Jan;85(1):27-32. doi: 10.2106/00004623-200301000-00005. PMID 12533568
- [Background] Kurtz S, Ong K, Lau E, Mowat F, Halpern M. Projections of primary and revision hip and knee arthroplasty in the United States from 2005 to 2030. J Bone Joint Surg Am. 2007 Apr;89(4):780-5. doi: 10.2106/JBJS.F.00222. PMID 17403800
- [Background] Schwartz AM, Farley KX, Guild GN, Bradbury TL Jr. Projections and Epidemiology of Revision Hip and Knee Arthroplasty in the United States to 2030. J Arthroplasty. 2020 Jun;35(6S):S79-S85. doi: 10.1016/j.arth.2020.02.030. Epub 2020 Feb 19. PMID 32151524